CLINICAL TRIAL: NCT01512732
Title: Validation of the Hebrew Version of the Montreal Affective Voices.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: HebVerMAV-HMO-CTIL
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Parkinson's Disease; Depression
MeSH Terms: conditions — Parkinson Disease; Depression

GROUPS / COHORTS (3):
- healthy control group: Young (20-49) and Older (50-70) healthy group (n=60)
- Parkinson's disease patients: (n=30).
- Major depressive disorder patients: (n=30).

SUMMARY:
Today, no non-verbal auditory stimuli that assess mental processing are available in Israel. The goal of this study is to make available a validated set of auditory stimuli in Israel. We created a computerized Hebrew version of the Montreal Affective Voices (MAV). The MAV is a novel tool for assessing mental processing. The MAV consists of 90 nonverbal affect bursts corresponding to nine different emotions (such as anger, fear, happiness etc.) recorded by ten different actors. The uniqueness of these affective bursts is that they do not contain verbal context, but rather express affective moods using the vowel /a/ (as in "apple"). In this study, the investigators will verify the new Hebrew version of MAV in healthy control groups. Next, the investigators will compare the mental processing ability in young vs. old population, using the MAV test. In addition, the investigators will assess mental processing in two pathologic study groups (Parkinson's disease, major depressive disorder) using the MAV test. The investigators intend to use the MAV tool in future research in Parkinson's disease and depression.

ELIGIBILITY:
Inclusion Criteria:

* Healthy group
* Parkinson's disease
* Major depressive disorder
* All participants will be competent and willing to give written informed consent. Patients over 65 and/or suspected to have a cognitive decline will be tested by the Mini-mental test and will be included in the study only if the score is above 26.

Exclusion Criteria:

* Non-competent or unable to give written informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy group, Parkinson's disease patients, Major depressive disorder patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-02

PRIMARY OUTCOMES:
Verifying the results achieved by Belin et al (2008) when using the Hebrew version of the MAV bursts in healthy control groups. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel